CLINICAL TRIAL: NCT02362932
Title: A Controlled Before and After Study to Measure the Effect of an Urban Sanitation Intervention on Child Health, in Low-income Neighborhoods of Maputo, Mozambique
Brief Title: The Effect of an Urban Sanitation Intervention on Child Health
Acronym: MapSan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 8345
Record Dates: First submitted 2015-02-04; First posted 2015-02-13 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2018-08

CONDITIONS: Diarrhea; Helminthiasis
MeSH Terms: conditions — Diarrhea; Helminthiasis | interventions — Sanitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Sanitation
  Interventions: Other: Sanitation
- Control (No Intervention): No sanitation

INTERVENTIONS:
Other: Sanitation — Shared sanitation
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine the health impact of a basic sanitation intervention in Maputo, Mozambique.

DETAILED DESCRIPTION:
We have designed a controlled, before-and-after (CBA) effectiveness study to estimate the health impacts of an urban sanitation intervention in informal neighborhoods of Maputo, Mozambique, including an assessment of whether exposures and health outcomes vary by localized population density. The intervention consists of private pour-flush latrines (to septic tank) shared by multiple households in compounds or household clusters. We will measure objective health outcomes in approximately 1000 children (500 children with household access to interventions, 500 controls using existing shared private latrines in poor sanitary conditions), at two time points: immediately before the intervention and at follow-up after 12 months. The primary outcome is combined prevalence of enteric infections among children under 5 years of age. Secondary outcome measures include soil transmitted helminth (STH) re-infection in children following baseline de-worming and prevalence of reported gastrointestinal illness. We will use exposure assessment, fecal source tracking, and microbial transmission modeling to examine whether and how routes of exposure for diarrheagenic pathogens and STHs vary and transmission impacts of the pathogens following introduction of effective sanitation. Our analysis will focus specifically on the impact of localized population density as a potential modifier of sanitation-related exposures.

ELIGIBILITY:
Inclusion Criteria:

* Children normally resident in households with access to new shared sanitation (the intervention) as selected by implementing organisation (WSUP) or control children normally resident in households sharing existing shared sanitation within geographically delimited project bounds and meeting WSUP site selection criteria (including number of people served)

Exclusion Criteria:

* Refusal to participate

Ages: 29 Days to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1866 (Actual)
Dates: Start 2015-02; Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Combined prevalence of bacterial and protozoan enteric infections | 12 month follow-up
  As identified via molecular assays on stool samples, we will measure combined prevalence of the following enteric infections: Campylobacter; Clostridium difficile, Toxin A/B; E. coli O157; Enterotoxigenic E. coli (ETEC) LT/ST; Shiga-like toxin producing E. coli (STEC) stx1/stx2; Salmonella; Shigella; Vibrio cholerae; Yersinia enterocolitica; Giardia; Cryptosporidium; and Entamoeba histolytica

SECONDARY OUTCOMES:
Combined helminth re-infection at 1 year following baseline de-worming | 12 month follow-up
  Combined prevalence of the following soil-transmitted helminths, as measured in stool samples via the Kato-Katz method: Ascaris spp., Trichuris spp., hookworm
Combined helminth re-infection at 1 year following baseline de-worming | 24 month follow-up
  Combined prevalence of the following soil-transmitted helminths, as measured in stool samples via the Kato-Katz method: Ascaris spp., Trichuris spp., hookworm
Period prevalence (7-day recall) of gastrointestinal illness | 12 month follow-up
  We will measure caregiver-reported symptoms of gastrointestinal illness, including diarrhea, vomiting, and abdominal pain.
Period prevalence (7-day recall) of gastrointestinal illness | 24 month follow-up
  We will measure caregiver-reported symptoms of gastrointestinal illness, including diarrhea, vomiting, and abdominal pain.
Height-for-age z-score | 24 month follow-up
  Height, measured by length/height boards, standardised to z-scores against WHO 2009 Child Growth Standards
Combined prevalence of bacterial and protozoan enteric infections | 24 month follow-up
  As identified via molecular assays on stool samples, we will measure combined prevalence of the following enteric infections: Campylobacter; Clostridium difficile, Toxin A/B; E. coli O157; Enterotoxigenic E. coli (ETEC) LT/ST; Shiga-like toxin producing E. coli (STEC) stx1/stx2; Salmonella; Shigella; Vibrio cholerae; Yersinia enterocolitica; Giardia; Cryptosporidium; and Entamoeba histolytica

CONTACTS AND LOCATIONS:
Overall Officials: Joe Brown, PhD, Principal Investigator — Georgia Institute of Technology (Georgia Tech); Oliver Cumming, MSc, Study Director — London School of Hygiene and Tropical Medicine
Locations (1):
- Health Research for Development, Maputo, Mozambique

REFERENCES:
- [Derived] Holcomb DA, Monteiro V, Capone D, Antonio V, Chiluvane M, Cumbane V, Ismael N, Knee J, Kowalsky E, Lai A, Linden Y, Mataveia E, Nala R, Rao G, Ribeiro J, Cumming O, Viegas E, Brown J. Long-term impacts of an urban sanitation intervention on enteric pathogens in children in Maputo city, Mozambique: study protocol for a cross-sectional follow-up to the Maputo Sanitation (MapSan) trial 5 years postintervention. BMJ Open. 2023 Jun 8;13(6):e067941. doi: 10.1136/bmjopen-2022-067941. PMID 37290945
- [Derived] Bick S, Buxton H, Chase RP, Ross I, Adriano Z, Capone D, Knee J, Brown J, Nala R, Cumming O, Dreibelbis R. Using path analysis to test theory of change: a quantitative process evaluation of the MapSan trial. BMC Public Health. 2021 Jul 16;21(1):1411. doi: 10.1186/s12889-021-11364-w. PMID 34271913
- [Derived] Knee J, Sumner T, Adriano Z, Anderson C, Bush F, Capone D, Casmo V, Holcomb D, Kolsky P, MacDougall A, Molotkova E, Braga JM, Russo C, Schmidt WP, Stewart J, Zambrana W, Zuin V, Nala R, Cumming O, Brown J. Effects of an urban sanitation intervention on childhood enteric infection and diarrhea in Maputo, Mozambique: A controlled before-and-after trial. Elife. 2021 Apr 9;10:e62278. doi: 10.7554/eLife.62278. PMID 33835026
- [Derived] Knee J, Sumner T, Adriano Z, Berendes D, de Bruijn E, Schmidt WP, Nala R, Cumming O, Brown J. Risk factors for childhood enteric infection in urban Maputo, Mozambique: A cross-sectional study. PLoS Negl Trop Dis. 2018 Nov 12;12(11):e0006956. doi: 10.1371/journal.pntd.0006956. eCollection 2018 Nov. PMID 30419034
- [Derived] Brown J, Cumming O, Bartram J, Cairncross S, Ensink J, Holcomb D, Knee J, Kolsky P, Liang K, Liang S, Nala R, Norman G, Rheingans R, Stewart J, Zavale O, Zuin V, Schmidt WP. A controlled, before-and-after trial of an urban sanitation intervention to reduce enteric infections in children: research protocol for the Maputo Sanitation (MapSan) study, Mozambique. BMJ Open. 2015 Jun 18;5(6):e008215. doi: 10.1136/bmjopen-2015-008215. PMID 26088809